CLINICAL TRIAL: NCT00538538
Title: Use of Subretinal Ranibizumab (Lucentis) in the Management of Submacular Hemorrhage in Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Subretinal Lucentis for Hemorrhagic Age-related Macular Degeneration (AMD)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This condition can now be managed in the office with an injection of Lucentis.
Sponsor: Corewell Health East (Other)
Responsible Party: Tarek Hassan, M.D., Associated Retinal Consultants, P.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC 2007-073
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Retinal Hemorrhage; Macular Degeneration
Keywords: Macular Degeneration; AMD; Hemorrhage; Wet AMD
MeSH Terms: conditions — Retinal Hemorrhage; Macular Degeneration; Hemorrhage | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Does not receive Gas bubble
  Interventions: Drug: vitrectomy with subretinal lucentis
- B (Active Comparator): Does receive gas bubble
  Interventions: Drug: vitrectomy with subretinal lucentis

INTERVENTIONS:
Drug: vitrectomy with subretinal lucentis — A gas bubble will be placed in the eye after the gel has been removed.
  Arms: B
Drug: vitrectomy with subretinal lucentis — These patients will have a vitrectomy where the gel is removed but will not receive the gas bubble.
  Arms: A

SUMMARY:
Visual outcomes of the eye with large subretinal hemorrhages (bleeding under the retina) due to Age-Related Macular Degeneration (AMD) are poor. The Submacular Surgery Trial (SST) showed that no statistically significant improvement in vision resulted from surgical removal of the layer of abnormal blood vessels causing the bleeding. However, placement of a gas bubble into the gel of the eye along with removal of the blood has shown some success. However, this does not treat the underlying condition of the AMD.

Intravitreal injections (into the gel of the eye) of a drug called Lucentis has been shown to be highly effective in the treatment of AMD, yet its penetration through areas of thick blood caused by subretinal hemorrhage is not known.

This study is proposing to treat the AMD causing the subretinal hemorrhage with a vitrectomy (surgery involving removing the gel inside the eye, and membrane layers of the eye) followed by Lucentis placed between the layers of the retina and then with or without a gas bubble.

In order to determine if the the subretinal Lucentis alone is beneficial, 5 of the 10 patients enrolled will get a gas bubble and the other 5 will not.

DETAILED DESCRIPTION:
Subjects will be followed for a period of 12 months. Based on photographs and other testing procedures, if it is deemed in the subject's best interest, the subject may receive monthly injections of Lucentis to help treat the AMD.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years
* Vision 20/200 or worse
* AMD with submacular hemorrhage
* Hemorrhage more than 25% of the lesion
* Fibrosis or scar not more than 25% of the entire lesion
* Hemorrhage less than 3 months old
* Vision loss occuring within 3 months

Exclusion Criteria:

* Pregnancy
* Participating in any other clinical trial
* Prior treatment for AMD
* Other medical conditions causing compromised vision
* Intraocular eye surgery within the previous 12 months
* Inability to obtain necessary eye photographs
* Systemic use of anti-VEGF agents
* Allergy to fluorescein dye
* Unable to complete all study visits
* Glaucoma filtering surgery
* Use of 2 or more treatments for glaucoma
* Lack of lens in the eye or absence of a posterior capsule

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of vitrectomy combined with a single dose of subretinal Ranibizumab (Lucentis - 0.5 mg) in patients with submacular hemorrhage and choroidal neovascular membranes secondary to AMD. | 12 months

SECONDARY OUTCOMES:
Mean change in visual acuity, angiographic area, retinal thickness by optical coherence tomography, mean number of retreatments required by 12 months. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Hassan, MD, Principal Investigator — Associated Retinal Consultants/William Beaumont Hosp.
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States